CLINICAL TRIAL: NCT05160870
Title: Genotype-phenotype Correlation and Pathogenic Mechanism in Hereditary Ataxia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: Wulab-sNfL in HA
Record Dates: First submitted 2021-12-06; First posted 2021-12-16 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2021-11

CONDITIONS: Hereditary Ataxia
MeSH Terms: conditions — Spinocerebellar Degenerations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators aimed to find appropriate biomarkers such as serum neurofilament light chain in reflecting disease severity in hereditary ataxia from a large cohort during long-term follow-up. The disease severity is indicated by clinical scales and brain MRI tests.

ELIGIBILITY:
Inclusion Criteria:

* genetically diagnosed as Spinocerebellar ataxia

Exclusion Criteria:

* deny follow-yp

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with Spinocerebellar ataxia
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-06-30 (Actual); Primary Completion 2022-12-25 (Estimated); Study Completion 2025-12-25 (Estimated)

PRIMARY OUTCOMES:
Serum neurofilament light chain | from 2021 to 2025
  Serum neurofilament light chain levels were collected among patients in preclinical or mild stage of Spinocerebellar ataxia, especially type 3.

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China